CLINICAL TRIAL: NCT04054310
Title: Non-Invasive Quantification of Liver Health in NASH (N-QUAN): A Prospective Diagnostic Accuracy Study
Brief Title: Non-Invasive Quantification of Liver Health in NASH (N-QUAN)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IIP137
Record Dates: First submitted 2019-08-05; First posted 2019-08-13 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Biopsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study-gate (Experimental): Single arm of biopsy naïve participants suspected of having NAFLD or NASH, who have been referred for a liver biopsy as part of routine clinical care
  Interventions: Diagnostic Test: Liver Multi Scan

INTERVENTIONS:
Diagnostic Test: Liver Multi Scan — MRI to create cT1, T2* and PDFF images of patients liver.
  Other Names: Biopsy

SUMMARY:
To evaluate, in patients with suspected NASH referred for liver biopsy, the diagnostic performance of CT1 at discriminating those with NAS≥4 & F≥2 from those without.

DETAILED DESCRIPTION:
NASH trials will often use the criteria proposed by the NASH Clinical Research Network (NASH-CRN), the NAS scoring system, to classify patients as suitable for study enrolment. NAS is a summation of the histology scores for fat (0-3), inflammation (0-3), and ballooning (0-2) with a score of 4 or 5 or higher regarded as NASH. Whilst the score doesn't include fibrosis, the rapidly evolving clinical trials landscape in NASH has seen a shift in emphasis from drugs proposed to target liver fat to the targeting of fibrosis. This was due to observations contrary to the previously held belief that fibrosis could not improve, and the data to support fibrosis being predictive of clinical outcomes. As a result, many clinical trials now require patients to have a NAS ≥4 or 5, with the regulatory accepted criteria requirement for at least a score of 1 for inflammation and 1 for ballooning, and evidence of fibrosis of stage 2 or more (scored using the Kleiner-Brunt (0-4) scale). The route by which a liver biopsy is indicated for inclusion to a clinical trial is usually based on patient presentation and clinical work-up. In the Primary care patient presents with clinical risk factors for NASH like metabolic syndrome. Blood biomarkers will be checked and if raised patient will be referred to the hepatology. In the secondary care patient might have a transient elastography and if CAP is equal or more than 280 and LSM is equal or more than 7 kPa, patient will have biopsy.

However clinical risk factors are often not sensitive enough, and NASH trials often suffer from high levels of screen fails at biopsy, meaning a large proportion are unnecessarily biopsied. Screening strategies are becoming increasingly more popular in order to reduce the number that fail screening and metrics derived from magnetic resonance imaging (MRI) such as T1-mapping and PDFF are emerging as promising diagnostic screening biomarkers in NASH.

MRI exploits the magnetic properties of hydrogen nuclei protons within a determined magnetic field. T1 mapping measures longitudinal relaxation time, a measure of how long it takes for protons to re-equilibrate their spins to the magnetic field after being excited by a radiofrequency pulse, and thus is an indicator of regional tissue water (proton) content. T1 mapping has shown promise as an effective biomarker of liver inflammation and fibrosis, as T1 relaxation time lengthens with increases in extracellular fluid (which may be caused by fibrosis and/or inflammation). The presence of iron however, which can be accurately measured from MRI-T2star (T2*) relaxation time, shortens the T1, and thus must be accounted for. An algorithm has been created (Perspectum Diagnostics) that allows for the bias introduced by elevated iron to be removed from the T1 measurements, yielding the iron corrected T1 (cT1). Iron corrected T1 (cT1) has been shown to correlate with fibro-inflammatory disease and can effectively stratify patients with NASH and cirrhosis (7).

MRI-PDFF is a ratio, expressed as a percentage, of the fraction of the MRI-visible protons attributable to fat divided by all MRI-visible protons in that region of the liver attributable to fat and water. Taking advantage of the chemical shift between fat and water, pulse sequences including fast spin echo and gradient-recalled echo (GRE) sequences can be used to acquire images at multiple echo times at which fat and water signals have different phases relative to each other. PDFF has been shown to have excellent correlation between histologically graded steatosis across the clinical range seen in NASH and high diagnostic accuracy in stratification of all grades of liver steatosis, although it is weaker in the presence of advanced fibrosis. Whilst PDFF does not correlate with other features of NASH, it has been reported that NAFLD patients with grade one steatosis are more likely to have characteristics of advanced liver disease such as fibrosis and ballooning, and changes in hepatic steatosis may be correlated with changes in other histological endpoints. Thus whilst some authors advise caution about using PDFF as a biomarker of NASH it has been well accepted by the NASH community as a biomarker for both enrolment and as an endpoint in NASH clinical trials (e.g. MOZART: NCT01766713; FLINT: NCT01265498).

Where cT1 appears to have an advantage over PDFF as a non-invasive biomarker for NASH, is in detection of patients with both disease activity (ballooning and inflammation) and fibrosis as cT1 has been reported to be correlated with ballooning, fibrosis and NAFLD activity score, and has been shown to predict clinical outcomes. As such it is emerging as a promising biomarker for both screening and as an endpoint in NASH clinical trials (NCT02421094; NCT02912260) particularly those investigating mechanisms of action of fibro-inflammation, or for distinguishing those with more advanced NASH with fibrosis. Both cT1 and PDFF can be acquired as part of the LiverMultiScan™ (LMS) imaging protocol (Perspectum Diagnostics Ltd, UK).

Based on the data reported in the literature, and from our preliminary analysis of N=109 biopsy-confirmed NAFL patients recruited from the two UK studies, both cT1 and PDFF appear to have potential to become diagnostic biomarkers, that may have utility for clinical trial population enrichment when used in conjunction with clinical risk factors. Specifically, for PDFF to identify participants who are more likely to have histopathologic findings of steatosis, and cT1 to identify participants who are more likely to have histopathologic findings of NASH, and NASH with fibrosis.

The primary objective of this study is to evaluate cT1 (Corrected T1) as a diagnostic biomarker that can be used, in conjunction with clinical risk factors, to identify patients who are more likely to have liver histopathologic findings of non-alcoholic steatohepatitis (NASH). Ideally, this biomarker should identify patients with a non-alcoholic fatty liver disease activity score (NAS) ≥ 4 and liver fibrosis (NASH/CRN Brunt/Kleiner scale) ≥ stage 2 on histopathologic assessment.

Based on our observations from earlier trials, our hypothesis is that we expect cT1 to have good diagnostic accuracy for discriminating those with NAS≥4 & F≥2 from those without

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects aged between 18 and 75 years old
* Ability to understand and sign a written informed consent forms
* Patients scheduled to undergo a standard of care diagnostic liver biopsy as follows
* Percutaneous biopsy with a 16 gauged needle passed into the right lobe
* Trans-jugular biopsy with an 18 gauged needle passed into the right lobe
* Patients who are suspected of having NAFLD, who are being considered for treatment, and presenting with two or more of the following risk factors for NASH
* Elevated liver enzymes (ALT≥40)
* BMI≥25kG/m^2
* Hypertension
* Type II diabetes
* Dyslipidameia
* Low High-density lipoprotein (HDL) (<40mg/dl in men or <50mg/dl in women)
* Hypertriglyceridemia (≥150mg/dl)
* Hypercholestrolemia (≥200mg/dl)
* Triglycerides (TG)/HDL>5.0

Exclusion Criteria:

* Prior histopathological diagnosis of NASH
* Inability to undergo a liver biopsy
* Prior or planned liver transplantation
* Patient scheduled to undergo a laparoscopic or wedge liver biopsy or biopsy taken from the left lobe
* Participation in an investigational new drug (IND) trial in the 30 days before enrolment
* Other known causes of chronic liver disease based on clinical criteria at the study site such as the following:
* Alcoholic liver disease
* Primary biliary cirrhosis
* Primary sclerosing cholangitis
* Autoimmune Hepatitis
* Wilson's disease, hemochromatosis, iron overload
* Alpha/1/Antitrypsin (A1AT) deficiency
* HCV, HBV
* History or diagnosis of cirrhosis and or hepatic decompensation including ascites, hepatic encephalopathy or variceal bleeding
* Clinically relevant drug or alcohol abuse within 12 months of screening
* Any contradiction or significant limitation to MRI scanning
* Claustrophobia preventing MR imaging (requires 15-30 minutes in scanning)
* Pacemaker or another implanted device
* Metal in body (such as an aneurysm clip) that might produce artefacts on abdominal MRI or might be adversely impacted by a high magnetic field
* Inability to lie flat, remain still or briefly hold breath as necessary during MR imaging
* Medical condition likely to produce significant hypervolemia like congestive heart failure
* Severe obesity complicating positioning in MR scanner
* Weight reduction surgery within 3 years
* Concomitant medical illnesses per investigators discretion (such as HIV infection, recent major surgery, uncontrolled heart disease, concurrent infection or fever of unknown origin, illicit drug use, cancer
* Clinically significant medical or psychiatric condition considered a high risk participation in an investigational study
* Failure to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of cT1 | 12 months
  To evaluate, in patients with suspected Nash referred for Liver biopsy, the diagnostic performance of cT1 at discriminating those patients with NAS≥4 & F≥2 from those patients without. In order to evaluate the diagnostic performance area under the receiver operative curve (AUROC) will be analysised.

SECONDARY OUTCOMES:
Diagnostics performance of PDFF | 12 months
  To evaluate, inpatients with suspected NASH referred for liver biopsy, the diagnostic performance of PDFF at discriminating those with NAS≥4 from those without, and those with Brunt Steatosis≥2 from those without. The diagnostic performance will be determined using area under the receiver operative curve (AUROC) analysis.
Correlation between cT1 and hisopathological features | 12 months
  To assess the correlation between cT1 and histopathological features of NASH and PDFF and histopathological features of NASH. The correlations will be explored using Spearman's Rho

CONTACTS AND LOCATIONS:
Overall Officials: Arun Sanyal, M.D., Principal Investigator — VCU School of Medicine
Locations (7):
- United States (7):
  - Arizona Liver Health, Chandler, Arizona
  - RUSH University Medical Center, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Liver Center of Texas, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Common wealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No